CLINICAL TRIAL: NCT04409743
Title: Harnessing Telehealth to Mitigate the Impact of the COVID-19 Pandemic on Sleep, Suicidality, and Neuropsychiatric Symptoms
Brief Title: Brief Telehealth CBT-I Intervention in the Context of the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-55940
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Sleep Disturbance; Insomnia
Keywords: Sleep; CBT-I; Cognitive Behavioral Therapy; COVID-19
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Active Comparator): The sleep treatment is Cognitive Behavioral Therapy for Insomnia (CBT-I). Participants randomized to this arm will begin treatment immediately after randomization.
  Interventions: Behavioral: Remote Cognitive Behavioral Therapy for Insomnia
- Waitlist (Other): The subjects assigned to the Waitlist condition will receive the same CBT-I treatment 7 months after randomization.
  Interventions: Behavioral: Remote Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Remote Cognitive Behavioral Therapy for Insomnia — Participants will meet with a psychologist through telehealth once a week for four weeks to complete a brief CBT-I intervention. Cognitive Behavioral Therapy for Insomnia consists of a cognitive therapy and a behavioral therapy. The cognitive therapy is designed to identify incorrect ideas about sleep, challenge their validity, and replace them with correct information. This therapy tries to reduce worry, anxiety, and fear that one won't sleep by providing accurate information about sleep. The behavioral therapy increases sleep quality by limiting excessive time spent in bed to increase homeostatic sleep drive and sleep consolidation.
  Other Names: CBT-I

SUMMARY:
The purpose of this study is to investigate whether an empirically validated treatment for insomnia (CBT-I) administered early in the course of sleep disturbance can prevent insomnia disorder or lessen negative mental health outcomes in the wake of the COVID-19 crisis in adults.

DETAILED DESCRIPTION:
The COVID-19 Pandemic and the resulting mass home confinement enacted to mitigate disease spread has created an environment of stress and drastic disruption to daily life. Increases in stress, social isolation, loss of daily routine, decreased physical activity, and excess screen time that are likely to arise as a function of the pandemic and mitigation efforts are risk factors for developing insomnia. Left unchecked, this acute insomnia can become chronic, resulting in increased risk of negative mental health outcomes such as depression, anxiety, and suicidality. The current proposal aims to test whether a telehealth intervention for insomnia can be used to not only prevent the progression of acute to chronic insomnia, but also prevent the worsening of neuropsychiatric symptoms, suicidality, and quality of life in those most vulnerable to negative mental health outcomes.

These aims will be achieved through a randomized 2-arm controlled trial design. 50 eligible adults experiencing sleep disturbances and who also have a history of depression and are in the at-risk group for COVID-19 will be randomized to receive either a sleep intervention (Cognitive Behavioral Therapy for Insomnia, CBT-I; n=25) or a 7-month waitlist (n=25). CBT-I improves sleep patterns through a combination of sleep restriction, stimulus control, mindfulness training, cognitive therapy targeting dysfunctional beliefs about sleep, and sleep hygiene education. Neuropsychiatric symptoms, Quality of Life, suicidality, and sleep disruption will be assessed at baseline (Week 0) and at the end of the sleep intervention (or Week 7) through online surveys and clinical interviews. Neuropsychiatric symptoms (anxiety and depression) and sleep disturbance (Insomnia Severity Index, and sleep diaries) will be assayed at baseline and each week throughout treatment/waitlist to assess week-to-week changes following an increasing number of CBT-I sessions. Neuropsychiatric symptoms, quality of life, suicidality, and sleep will be assessed again at 3-months, 7-months, and 13-months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Access to the internet
* Subjective complaint of sleep disturbance (ISI ≥10) that began after March 1, 2020 or the COVID-19 Pandemic (self-reported during DUKE Interview)
* Lives in the United States

Exclusion Criteria:

* Presence of suicidal ideation representing high risk as measured by the Sheehan-Suicide Tracking Scale (S-STS).
* Use of medication specifically prescribed for sleep disturbance and unwilling or unable to discontinue more than one week prior to baseline data collection.
* Current or lifetime history of bipolar disorder or psychosis
* Current substance abuse or dependence
* Not able to verbalize understanding of involvement in research and provide written, informed consent
* Not fluent or literate in English
* Unstable pharmacotherapy for other mental health disorders
* Severe impediment to vision, hearing, and/or hand movement, likely to interfere with the ability to complete assessments, or are unable and/or unlikely to follow study protocols
* Working rotating shift that overlaps with 2400h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Clinical Diagnosis Over Time | Assessed at week 0, month 3, month 7, and month 13
  Whether the participant has an insomnia clinical diagnosis will be measured by the DUKE. The DUKE is a structured interview which screens for sleep disorders in accordance with criteria of both the DSM-IV and the international classification of sleep disorders (ICSD-2). The DUKE is composed of 4 modules that assess sleep disorder symptoms associated with complaints of insomnia, sleep disorders associated with complaints of hypersomnia, circadian rhythm sleep disorders, and sleep disorders associated with parasomnias.
Change in Patient Health Questionnaire-9 (PHQ-9) Scale Score as a Measure of Depression Symptoms Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  The PHQ-9 is a self-administered 9-item 0 to 3 scale (0 = not at all, 3 = nearly every day) questionnaire that assess each of the 9 DSM-IV depression criteria. The total score ranges from 1 - 27 which measures the severity of the reported depression with consideration for both Major Depressive Disorder and other depressive disorders based on the number of items that were rated a 2 to 3.
Change in Generalized Anxiety Disorder-7 (GAD-7) Scale Score Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  The GAD-7 is a widely used diagnostic self- report scale that screens, diagnoses, and assess severity of anxiety disorder. The GAD-7 is a 7-item 0 to 3 (0 = Not at all, 3 = Nearly every day) scale that measures the degree of severity of anxiety over the last 2 weeks with a total score ranging from 0 to 21, with a higher score indicating a more severe anxiety.
Change in Insomnia Severity Index (ISI) Scale Score Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  Subjective ratings of sleep disturbance and insomnia severity will be assessed with the Insomnia Severity Index. The Insomnia Severity Index (ISI) is a 7-item self-report measure of insomnia type, severity, and impact on functioning. The items consist of severity of sleep onset, sleep maintenance, early morning awakenings, sleep dissatisfaction, interference with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Items are scored from 0 to 4 (0 = no problem, 4 = very severe problem). Score ranges of insomnia are: 0-7 absent, 8-14 sub-threshold, 15-21 moderate, and 22-28 severe. The ISI has good validity and reliability.
Change in Quality of Life (SF-36) Scale Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  The SF-36 is a 36-item self-administered survey to assess comprehensive quality-of-life measures. It consists of eight sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, and mental health. This survey is widely used and has been proven to be a reliable indicator of quality-of-life measures. The global score range is 0-100, with higher scores indicating better health conditions.
Change in Sheehan Suicidality Tracking Scale (S-STS) Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  Suicidality ideation and behaviors will be measured by the S-STS. The S-STS is a 16-item 0 to 4 scale (0 = no problem, 4 = very severe problem) that assesses the risk of suicidality. For this outcome measure, 15 items (excluding #13) are summed for an overall score range of 0 to 45 (higher scores indicate more severe problems).
Change in UCLA Loneliness Scale Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  Loneliness risk factors will be assessed with the UCLA Loneliness Scale that measures a participant's subjective feelings of loneliness and social isolation. The UCLA Loneliness Scale has 20 items, each on a 1 to 4 scale (1 = Never, 4 = Often), summed for an overall range of 20 to 80 with higher scores indicating greater degrees of loneliness.
Change in Social Network Index (SNI) Scale Score Over Time | Assessed at week 0, month 7, and month 13
  The Social Network Index is a 12-item questionnaire that assess participation in different types of social relationships. The 12 types of relationships (e.g. friend, children, spouse, religious group member) are scored by the number network members they communicate with at least every 2 weeks.
Change in Perceived Stress Scale Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  The Perceived Stress Scale is a widely used self-reported questionnaire that assesses how stressful participants believe their live is. Items are generalized and measure the degree participants judge their lives to be uncontrollable and unpredictable over the course of the previous month.
Change in Screen Time- Self Report Over Time | Assessed at week 0, week 7, month 3, month 7, and month 13
  Self-report questions regarding screen time will be included in the Coronavirus Health Impact Survey. Questions measure the amount of time spent per day, over the course of the two most recent weeks, using an electronic device.
Change in International Physical Activity Questionnaire (IPAQ) Scale Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  The International Physical Activity Questionnaire assess an individual's physical activity across 5 life domains over the last 7 days. The activity domains consist of physical activity related to work, transportation, housework and caring for family, and recreation and sports as well as the amount of time spent sitting. The IPAQ has high reliability and validity and has been widely used to measure comparable estimates of physical activity in large populations.

SECONDARY OUTCOMES:
Change in Sleep Onset Latency (SOL) as a Measure of Sleep Continuity Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  Sleep Onset Latency (SOL) is the time (minutes) from "lights out" to actually falling asleep (sleep onset) based on sleep logs.
Change in Number of Awakenings as a Measure of Sleep Continuity Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  Number of Awakenings is determined by number of times of awakening as reported on sleep logs.
Change in Wake After Sleep Onset (WASO) as a Measure of Sleep Continuity Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  Wake After Sleep Onset (WASO) are periods of wakefulness occurring after sleep onset, before final awakening (sleep offset).
Change in Total Sleep Time (TST) as a Measure of Sleep Continuity Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  Total Sleep Time (TST) is the total time spent asleep, from the start of sleep onset to sleep offset subtracting any periods of wakefulness.
Change in Sleep Efficiency (SE) as a Measure of Sleep Continuity Over Time | Assessed at week 0, weekly from weeks 2 to 7, month 3, month 7, and month 13
  Sleep Efficiency (SE) is calculated as TST divided by total time spent in bed, multiplied by 100.
Change in Beck Depression Inventory-II (BDI) Scale Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  This measure is of the Beck Depression Inventory-II total score after excluding one sleep item. The average item score for the remaining 20 items will be multiplied by 21 (the original number of items), to create a modified depression scale that maintains the original range (ranges: 0-13 minimal, 14-19 mild, 20-28 moderate, and 29-63 severe).
  The BDI-II is a 21-item self-report scale with high validity and reliability that assesses the severity of depression symptoms. The depression items consist of: sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping pattern, irritability, changes in appetite, concentration difficulty, tiredness or fatigue, and loss of interest in sex. Items are scored from 0 to 3, and higher scores indicate greater levels of severity.
Change in Beck Anxiety Inventory (BAI) Scale Score Over Time | Assessed at week 0, month 3, month 7, and month 13
  Clinical anxiety symptoms will be measured by the BAI. The BAI is a 21-item self-report scale that assesses the severity of anxiety symptoms. Items are scored from 0 to 3 (0 = not at all, 3 = severe). Higher scores indicate greater levels of severity, and the ranges for anxiety levels are: 0-9 normal to minimal, 10-18 mild to moderate, 19-29 moderate to severe, and 30-63 severe. The BAI consists of two factors: somatic and cognitive.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Goldstein-Piekarski, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] O'Hora KP, Osorno RA, Sadeghi-Bahmani D, Lopez M, Morehouse A, Kim JP, Manber R, Goldstein-Piekarski AN. Viability of an Early Sleep Intervention to Mitigate Poor Sleep and Improve Well-being in the COVID-19 Pandemic: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2022 Mar 14;11(3):e34409. doi: 10.2196/34409. PMID 34995204